CLINICAL TRIAL: NCT07062510
Title: The Effects of Balanced Seating Pressure on Pelvic Asymmetry in Under-Buttocks Pressure, Spinal Alignment, and Lower Back Pain: A Pilot Study
Brief Title: The Effects of Balanced Seating Pressure on Pelvic Asymmetry: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2303070089
Record Dates: First submitted 2025-06-22; First posted 2025-07-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-06

CONDITIONS: Lower Back Pain; Scoliosis Patients
Keywords: sitting pressure; Under-Buttocks Pressure; Dasuit; Pelvic asymmetry; Spinal alignment deviation (SAD)
MeSH Terms: conditions — Low Back Pain | interventions — WASH protein, Drosophila

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dasuit to Placebo (Other): This group of patients will first undergo Dasuit intervention then Placebo intervention
  Interventions: Device: Dasuit Cusion; Device: Placebo; Other: Washout
- Placebo to Dasuit (Other): This group of patients will first undergo Placebo intervention then Dasuit intervention
  Interventions: Device: Dasuit Cusion; Device: Placebo; Other: Washout

INTERVENTIONS:
Device: Dasuit Cusion — The Dasuit cushion is placed on a 40X40X40 wooden box as a chair, and the pressure seating mat is placed on the cushion. Participants were asked to sit on the cushion with hips, knees, and ankles positioned at approximately 90° angles at ease. A tablet was mounted in front of the chair at 30-40 cm from the eyes and at a downward viewing angle of 5-10 degrees. Participants were instructed to watch a 10-minute video to maintain a fixed gaze and minimize head movement. The patient was to sit on the cushion at ease for 1 minute to adjust to the cushion, then under-buttock pressure was recorded for 10 mins.
Device: Placebo — The placebo cushion is placed on a 40X40X40 wooden box as a chair, and the pressure seating mat is placed on the cushion. Participants were asked to sit on the cushion with hips, knees, and ankles positioned at approximately 90° angles at ease. A tablet was mounted in front of the chair at 30-40 cm from the eyes and at a downward viewing angle of 5-10 degrees. Participants were instructed to watch a 10-minute video to maintain a fixed gaze and minimize head movement. The patient was to sit on the cushion at ease for 1 minute to adjust to the cushion, then under-buttock pressure was recorded for 10 mins.
Other: Washout — A 10 min washout period is in between the two interventions. The paitent is asked to walk around at ease.

SUMMARY:
The goal of this clinical trial is to learn if the DaSuit® cushion helps reduce discomfort caused by sitting in adults with non-specific low back pain. It will also assess the safety and physical effects of using the DaSuit® cushion. The main questions it aims to answer are:

1. Does the DaSuit® cushion distribute the pressure evenly on both under-buttock pressure compared to a placebo cushion?
2. Does the DaSuit® cushion improve spinal alignment compared to a placebo cushion?
3. What discomfort or adverse events do participants experience when using the DaSuit® cushion?

Researchers will compare the DaSuit® cushion to a placebo cushion (a look-alike cushion without therapeutic effect) to see if the DaSuit® cushion works to relieve sitting-induced discomfort.

Participants will:

1. Use the DaSuit® cushion or a placebo cushion in a randomized order, with each sitting session lasting 10 minutes
2. Complete both conditions with a 10-minute washout period between sessions
3. Sit on a standardized wooden chair with a pressure sensor mat placed on the cushion surface
4. Keep a fixed posture with hips, knees, and ankles at approximately 90 degrees
5. Watch a 10-minute video on a tablet positioned 30-40 cm in front of them at a 5-10 degree downward angle to maintain a steady gaze
6. Undergo spinal imaging immediately after each session, maintaining the same seated posture
7. Report any discomfort or pain experienced during or after each session

DETAILED DESCRIPTION:
Trial Design This study is designed as a randomized, double-blind, placebo-controlled, two-period crossover trial to be conducted at the Department of Rehabilitation, Taoyuan Chang Gung Memorial Hospital. A total of 24 participants will be screened, with an estimated 20 completing the full protocol. Participants will be randomly assigned to one of two treatment sequences: Group A will receive the DaSuit® cushion followed by the placebo cushion; Group B will receive the placebo cushion followed by the DaSuit® cushion. Each intervention period will last approximately 10 minutes, separated by a 10-minute washout interval to minimize potential carry-over effects. The crossover design is chosen to reduce between-subject variability, as each participant will serve as their own control.

Participants The study will not involve patients or the public in the design, conduct, reporting, or dissemination.

Inclusion criteria are as follows: (1) adults aged 20 to 50 years; (2) experiencing non-specific low back pain exacerbated by sitting, with a VAS score between 3 and 7; (3) height between 150-180 cm; (4) BMI between 18.5-24; and (5) radiographically verified hemi-pelvic height discrepancy ≥ 0.5 cm in a seated posture.

Exclusion criteria include: (1) inability to sit for 20 minutes; (2) MMSE < 24; (3) significant spinal or pelvic disorders (e.g., fractures, prior surgeries, herniated discs with nerve compression); (4) diagnosed scoliosis with a Cobb angle ≥ 20°; (5) recent use of analgesics or muscle relaxants; (6) pregnancy; and (7) skin conditions affecting sitting tolerance. All participants will provide written informed consent following clinical pelvic examination confirming asymmetry.

Interventions Each participant will undergo both intervention conditions in a randomized order. In each session, the participant will sit for 10 minutes on either the DaSuit® cushion or the placebo cushion, placed on a standardized 40×40×40 cm wooden chair. A pressure sensor mat will be placed on the cushion surface to measure under-buttock pressure. Following the sitting period, pain intensity will be assessed using the VAS, and an anterior-posterior full-spine X-ray will be taken. After a 10-minute washout period-during which the participant will be instructed to walk-the alternate cushion condition will be administered.

Outcome Measures Adverse events will be monitored throughout the study. Participants will be asked to report any discomfort or pain during or after each session. No adverse events are expected.

Primary outcomes include:

Under-buttock pressure:

* X and Y coordinates of center of force
* Total force applied to the cushion
* Area of force distribution
* Maximum pressure (mmHg)
* Area exceeding a defined percentage of maximum pressure
* Right/Left peak pressures
* Distance from center of force to Right/Left peak pressure points

Spinal alignment parameters:

* Spinal alignment deviation (SAD; C7-S1) Participants will again sit upright on the test chair without a cushion, and a frontal full-spine radiograph will be taken. The deviation will be calculated as the horizontal distance between the vertical lines passing through the center of the seventh cervical vertebra (C7 plumb line) and the center of the first sacral vertebra (S1 plumb line). This measurement reflects the lateral displacement of the spine and serves as an indicator of coronal imbalance.
* Pelvic height discrepancy (PHD) Pelvic height discrepancy (PHD) will be determined by measuring the vertical distance between the highest point of the iliac crest and the lowest point of the ischial tuberosity on both sides. A side-to-side difference of ≥0.5 cm will be used as the diagnostic threshold for pelvic asymmetry.
* Shoulder height discrepancy (SHD) While shoulder height discrepancy (SHD) is listed as a secondary outcome, its assessment will be based on the vertical difference between the acromion landmarks on both sides, if visible within the imaging field.

Pain intensity, measured via the visual analog scale (VAS)

Instrumentation and Procedures Pressure Mapping and Sitting Protocol: The cushion will be positioned on a 40×40×40 cm wooden box serving as a chair, with a pressure mat placed on top. Participants will sit with hips, knees, and ankles at approximately 90° angles. A tablet will be mounted at 30-40 cm distance and a downward viewing angle of 5-10° to maintain visual focus and reduce head movement. Participants will sit for one minute to acclimate, after which under-buttock pressure will be recorded continuously for 10 minutes.

Radiographic Procedure: For spinal imaging, the chair will be placed on a 20 cm X-ray platform. A 40×40×20 cm footrest will ensure consistent lower limb positioning during imaging. The imaging field will extend from the external auditory meatus to the seat base. Participants will maintain a natural sitting posture for 10 seconds prior to image capture.

Randomization and Blinding Randomization will be performed using a computer-generated sequence with a 1:1 allocation ratio. The sequence will be prepared by an independent statistician not involved in recruitment or data collection. Allocation concealment will be achieved through the use of sequentially numbered, opaque, sealed envelopes (SNOSE), managed by staff independent of the enrollment process. Both the DaSuit® and placebo cushions are designed to be visually indistinguishable. Participants will be blinded to the cushion type. However, due to logistical constraints, outcome assessors will not be blinded.

Statistical Analysis As a pilot study, the primary objective is to assess feasibility and obtain preliminary effect estimates for planning future trials. The sample size is not based on formal power calculations and results should be interpreted with caution regarding external validity.

Within-subject comparisons between the DaSuit and placebo conditions will be analyzed using paired t-tests. To examine potential sequence effects, between-group comparisons (Group A vs. Group B) will be conducted using independent t-tests. A two-tailed p-value of < 0.05 will be considered statistically significant.

All analyses will use complete case data; missing data are not anticipated. If missingness exceeds 10% in future trials, per-protocol analysis will serve as the primary strategy, supplemented by sensitivity analyses as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. adults aged 20 to 50 years
2. adults had low back pain non-specific but exacerbated by sitting with VAS score between 3-7
3. body height between 150-180 cm
4. BMI between 18.5-24
5. a radiographically verified hemi-pelvic height discrepancy of ≥ 0.3 cm in sitting posture
6. willing to participate and cooperate throughout the whole intervention session

Exclusion Criteria:

1. inability to sit for 20 minutes
2. MMSE < 24
3. significant spinal/pelvic disorders (e.g., fractures, surgeries, herniated discs with nerve compression)
4. scoliosis with Cobb angle ≥ 20°
5. recent use of pain killers and/or muscle relaxants
6. pregnancy
7. skin conditions affecting sitting tolerance.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Pelvic height discrepancy (PHD) | Periprocedural
  Measurement of the distance between the horizontal lines at the highest points of the bilateral iliac crests on the post-intervention whole spine radiographic imaging.
Right and Left peak pressures | Periprocedural
  This study will utilize the Sensing Tex® Seating Mat Dev Kit 1.9, a high-resolution textile-based pressure sensing system. The mat consists of a 16 × 16 matrix of 256 round sensor elements with a spatial resolution of 20 mm, embedded in a flexible textile structure. It is designed to be non-intrusive and can be placed directly between the seat surface and the participant without affecting comfort or posture.
  Right and left peak pressure values are determined by identifying the highest recorded pressure within the respective right and left hemispheres of the sensing matrix, defined relative to the midline axis of the mat. This bilateral analysis enables precise quantification of side-to-side pressure imbalance.

SECONDARY OUTCOMES:
Shoulder height discrepancy | Periprocedural
  The vertical distance between horizontal lines drawn along the superior borders of the clavicles on the radiograph.
Spinal alignment deviation | Periprocedural
  Measurement of the distance between the central C7 plumb line and the central S1 plumb line on an anteroposterior spinal radiograph.
X and Y coordinates of the center of pressure (mmHg) and Right/Left peak pressures | Periprocedural
  This study will utilize the Sensing Tex® Seating Mat Dev Kit 1.9, a high-resolution textile-based pressure sensing system. The mat consists of a 16 × 16 matrix of 256 round sensor elements with a spatial resolution of 20 mm, embedded in a flexible textile structure. It is designed to be non-intrusive and can be placed directly between the seat surface and the participant without affecting comfort or posture.
  X and Y coordinates of the center of pressure (mmHg) and Right/Left peak pressures
Total contact area | Periprocedural
  This study will utilize the Sensing Tex® Seating Mat Dev Kit 1.9, a high-resolution textile-based pressure sensing system. The mat consists of a 16 × 16 matrix of 256 round sensor elements with a spatial resolution of 20 mm, embedded in a flexible textile structure. It is designed to be non-intrusive and can be placed directly between the seat surface and the participant without affecting comfort or posture.
  The total contact area is measured by the number of sensors whose readings are above 0.
Area of values above 75% of the peak pressure | Periprocedural
  This study will utilize the Sensing Tex® Seating Mat Dev Kit 1.9, a high-resolution textile-based pressure sensing system. The mat consists of a 16 × 16 matrix of 256 round sensor elements with a spatial resolution of 20 mm, embedded in a flexible textile structure. It is designed to be non-intrusive and can be placed directly between the seat surface and the participant without affecting comfort or posture.
  Of the overall area, we count the senors whose values are above 75% of the peak pressure measured overall
Visual Analog Pain Scale | Periprocedural
  The Visual Analogue Scale (VAS) is a simple tool used in clinical and research settings to measure subjective experiences such as pain.
  It typically consists of a 10-cm horizontal line anchored by two extremes (e.g., "no pain" to "worst pain imaginable"), and participants mark a point along the line that best represents their current intensity of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Cheng Pei, M.D, PhD., Study Director — Chang Gung Memorial Hospital
Locations (1):
- Taoyuan Chang Gung Memorial Hospital, Taoyuan District, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including pressure sensor outputs, pelvic/spinal alignment measurements, and pain scores, will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 12 months post-publication and available for 3 years.
Access Criteria: Available to qualified investigators for academic use upon approval of a research proposal and signed data-sharing agreement.